CLINICAL TRIAL: NCT00617604
Title: Efficacy and Safety of Alefacept in Combination With Tacrolimus, Mycophenolate Mofetil and Steroids in de Novo Kidney Transplantation - a Multicenter, Randomized, Double-Blind, Placebo Controlled, Parallel Group Study
Brief Title: A Study to Assess the Efficacy and Safety of Alefacept in Kidney Transplant Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0485-CL-E201; 2007-002092-14 (EudraCT Number)
Record Dates: First submitted 2008-02-06; First posted 2008-02-18 (Estimated); Results first posted 2016-02-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-01

CONDITIONS: De Novo Kidney Transplantation
Keywords: kidney transplant; alefacept
MeSH Terms: interventions — Alefacept; Tacrolimus; Mycophenolic Acid; Steroids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo administered intra-operatively as an intravenous (IV) bolus on Day 0, another IV bolus on Day 3 and weekly subcutaneous injections thereafter for 12 weeks. Participants also received tacrolimus, mycophenolate mofetil (MMF) and steroid treatment.
  Interventions: Drug: placebo; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Drug: Steroids
- Alefacept (Experimental): Participants received 7.5 mg alefacept administered intra-operatively as an IV bolus on Day 0, another 7.5 mg IV bolus on Day 3, and weekly subcutaneous injections of 15 mg alefacept thereafter for 12 weeks. Participants also received tacrolimus, MMF and steroid treatment.
  Interventions: Drug: Alefacept; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Drug: Steroids

INTERVENTIONS:
Drug: Alefacept — IV and subcutaneous injection
  Other Names: Amevive
  Arms: Alefacept
Drug: placebo — IV and subcutaneous injection
  Arms: Placebo
Drug: Tacrolimus — The initial daily dose was 0.2 mg/kg orally given in 2 doses commencing 24 hours after completion of surgery.
Drug: Mycophenolate Mofetil — Mycophenolic mofetil was administered as 750 mg twice per day orally
Drug: Steroids — Methylprednisolone or equivalent:
  Day 0: 500 - 1000 mg IV bolus Day 1: 125 - 250 mg IV bolus
  Prednisone or equivalent:
  Days 2 - 14: 20 - 30 mg orally Days 15 - 28: 10 - 20 mg orally Days 29 - 60: 10 - 15 mg orally Days 61 onwards: 5 - 10 mg orally

SUMMARY:
The purpose of this study is to determine whether alefacept is effective and well tolerated when used with a combination of tacrolimus, mycophenolate mofetil and steroids versus a combination therapy of placebo, tacrolimus and steroids in the prevention of kidney transplant rejection.

ELIGIBILITY:
Inclusion Criteria:

* Subject with end stage kidney disease who is a suitable candidate for primary kidney transplantation or retransplantation
* Male or female subject at least 18 years of age and younger than 65 years
* Subject receiving a kidney transplant from a non-human leucocyte antigen (HLA) identical living donor or deceased HLA identical/non-HLA identical donor between 5 and 59 years of age with compatible ABO blood type (Blood group system A, B, AB and 0)

Exclusion Criteria:

* Subject has a panel reactivity antibody grade > 20% in the previous 6 months and/or had had a previous graft survival shorter than 1 year due to immunological reasons
* Subject received a kidney transplant from a non-heart beating donor
* Subject has received a kidney transplant from a 50 - 59 year old donor with two of the following three factors: history of hypertension, cerebrovascular accident as cause of death, final pre-procurement serum creatinine > 1.5 mg/dL (united network for organ sharing [UNOS] expanded criteria donor)
* Cold ischemia time of the donor kidney is ≥ 30 hours

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 218 (Actual)
Dates: Start 2007-12; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Europe B.V.
Locations (32):
- Vienna, Austria
- Belgium (4):
  - Brussels
  - Ghent
  - Leuven
  - Liège
- Prague, Czechia
- France (7):
  - Créteil
  - Le Kremlin-Bicêtre
  - Montpellier
  - Nantes
  - Nice
  - Paris
  - Toulouse
- Germany (2):
  - Bochum
  - Regensburg
- Budapest, Hungary
- Italy (4):
  - Bologna
  - Padua
  - Rome
  - Siena
- Maastricht, Netherlands
- Poland (3):
  - Bydgoszcz
  - Poznan
  - Szczecin
- Spain (5):
  - Barcelona
  - Llobregat
  - Madrid
  - Málaga
  - Santander
- Sweden (2):
  - Gothenburg
  - Uppsala
- Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 221 patients screened, 218 patients were enrolled into the study at 30 centers across 12 countries.
Period: Overall Study
Arm/Group | Placebo | Alefacept
Started | 110 | 108
Received Treatment | 107 | 105
Completed 12 Weeks of Treatment | 89 | 83
Completed | 92 (Completed Month 6 assessment) | 88 (Completed Month 6 assessment)
Not Completed | 18 | 20
Not completed — Death | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Miscellaneous Reasons | 8 | 10
Not completed — Withdrawal by Subject | 4 | 6
Not completed — Randomized but Never Received Study Drug | 3 | 3

BASELINE CHARACTERISTICS:
Population: All randomized patients who took at least 1 dose of study drug (Safety Analysis Set).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Alefacept | Total
Number analyzed (Participants) | 107 | 105 | 212
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (11.3) | 44.2 (11.9) | 45.4 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 40 | 73
  Male | 74 | 65 | 139

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Biopsy-confirmed Acute T-cell Mediated Rejection at Month 6 Assessed by Local Review
Description: Biopsies were graded by the clinical site pathologist.according to the Banff 97/05 updated histological classification:
  * Grade IA: significant interstitial infiltration (>25% parenchyma affected) and foci of moderate tubulitis;
  * Grade IB: significant interstitial infiltration (>25% parenchyma affected) and foci of severe tubulitis;
  * Grade IIA: mild to moderate intimal arteritis;
  * Grade IIB: severe intimal arteritis comprising >25% of the luminal area;
  * Grade III: "transmural" arteritis and/or arterial fibrinoid change and necrosis of medial smooth muscle cells with accompanying lymphocyte inflammation.
  A biopsy confirmed acute rejection was an event of suspected acute rejection confirmed by a graft biopsy result of Banff grade ≥ 1.
  The Kaplan-Meier estimate of biopsy-confirmed acute T-cell mediated rejection within the first 6 months following transplantation is reported. Participants lost to follow-up or with missing outcomes were censored at their last follow up visit.
Time Frame: 6 months
Population: Full analysis set (all randomized and transplanted participants who received at least 1 dose of study drug)
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Alefacept
Number analyzed (Participants) | 107 | 105
percentage of participants | 6.7 [2.7 to 10.7] | 10.6 [5.6 to 15.6]
Statistical Analysis 1: Comparison: Placebo vs Alefacept; Test type: Superiority or Other; Difference = 3.9, 90% CI 2-sided [-2.5 to 10.3]

2. Secondary Outcome: Percentage of Participants With Biopsy Confirmed Antibody-Mediated Acute Rejection at Month 6
Description: Biopsies were graded by the clinical site pathologist.according to the Banff 97/05 updated histological classification:
  Acute antibody-mediated rejection - documented anti-donor antibody ('suspicious for' if antibody not demonstrated):
  * Grade I: acute tubular necrosis-like - complement split product positive (C4d+), minimal inflammation;
  * Grade II: capillary-margination and/or thromboses, C4d+
  * Grade III: arterial - v3, C4d+.
  A biopsy confirmed acute rejection was an event of suspected acute rejection confirmed by a graft biopsy result of Banff grade ≥ 1.
  The Kaplan-Meier estimate of biopsy-confirmed antibody-mediated acute rejection within the first 6 months following transplantation is reported. Participants lost to follow-up or with missing outcomes were censored at their last follow up visit.
Time Frame: 6 months
Population: Full analysis set
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Alefacept
Number analyzed (Participants) | 107 | 105
percentage of participants | 2.9 [0.2 to 5.5] | 3.8 [0.7 to 6.9]
Statistical Analysis 1: Comparison: Placebo vs Alefacept; Test type: Superiority or Other; Difference = 1.0, 90% CI 2-sided [-3.1 to 5.0]

3. Secondary Outcome: Percentage of Participants With Biopsy Confirmed Acute Rejection (T-Cell Mediated or Antibody Mediated) at Month 6
Description: Biopsies were graded by the clinical site pathologist.according to the Banff 97/05 updated histological classification. A biopsy confirmed acute rejection was an event of suspected acute rejection confirmed by a graft biopsy result of Banff grade ≥ 1.
  The Kaplan-Meier estimate of biopsy-confirmed acute T-cell mediated or antibody-mediated rejection within the first 6 months following transplantation is reported. Participants lost to follow-up or with missing outcomes were censored at their last follow up visit.
Time Frame: 6 months
Population: Full analysis set
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Alefacept
Number analyzed (Participants) | 107 | 105
percentage of participants | 9.3 [4.7 to 14.0] | 12.4 [7.1 to 17.7]
Statistical Analysis 1: Comparison: Placebo vs Alefacept; Test type: Superiority or Other; Difference = 3.0, 90% CI 2-sided [-4.0 to 10.1]

4. Secondary Outcome: Percentage of Participants With Biopsy Confirmed Acute Mixed T-Cell Mediated and Antibody-Mediated Rejection at Month 6
Description: Biopsies were graded by the clinical site pathologist.according to the Banff 97/05 updated histological classification. A biopsy confirmed acute rejection was an event of suspected acute rejection confirmed by a graft biopsy result of Banff grade ≥ 1.
  The Kaplan-Meier estimate of biopsy-confirmed acute mixed T-cell mediated and antibody-mediated rejections within the first 6 months following transplantation is reported. Participants lost to follow-up or with missing outcomes were censored at their last follow up visit.
Time Frame: 6 months
Population: Full analysis set
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Alefacept
Number analyzed (Participants) | 107 | 105
percentage of participants | 0.0 [0.0 to 0.0] | 1.0 [0.0 to 2.5]
Statistical Analysis 1: Comparison: Placebo vs Alefacept; Test type: Superiority or Other; Difference = 1.0, 90% CI 2-sided [-0.6 to 2.5]

5. Secondary Outcome: Percentage of Participants With Acute Rejection Diagnosed by Signs and Symptoms at Month 6
Description: Acute rejection diagnosed by signs and symptoms, including biopsy-confirmed or suspected (not confirmed by biopsy - i.e. no biopsy was performed or biopsy did not confirm an acute T-cell mediated rejection). The Kaplan-Meier estimate of acute rejection diagnosed by signs and symptoms within the first 6 months following transplantation is reported. Participants lost to follow-up or with missing outcomes were censored at their last follow up visit.
Time Frame: 6 months
Population: Full analysis set
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Alefacept
Number analyzed (Participants) | 107 | 105
percentage of participants | 27.4 [20.3 to 34.6] | 22.3 [15.6 to 29.1]
Statistical Analysis 1: Comparison: Placebo vs Alefacept; Test type: Superiority or Other; Difference = -5.1, 90% CI 2-sided [-14.9 to 4.7]

6. Secondary Outcome: Percentage of Participants With Clinically Treated Acute Rejection at Month 6
Description: Patients who received immunosuppressive medications for the treatment of suspected or biopsy-confirmed acute rejections were considered to have a clinically-treated acute rejection. The Kaplan-Meier estimate of clinically treated acute rejection within the first 6 months following transplantation is reported. Participants lost to follow-up or with missing outcomes were censored at their last follow-up visit.
Time Frame: 6 months
Population: Full analysis set
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Alefacept
Number analyzed (Participants) | 107 | 105
percentage of participants | 24.8 [17.9 to 31.7] | 15.4 [9.6 to 21.2]
Statistical Analysis 1: Comparison: Placebo vs Alefacept; Test type: Superiority or Other; Difference = -9.4, 90% CI 2-sided [-18.5 to 0.0]

7. Secondary Outcome: Percentage of Participants With Steroid-resistant Acute Rejection at Month 6
Description: A steroid-resistant acute rejection is defined as a rejection episode which did not resolve following treatment with corticosteroids. In the case that a rejection episode was not treated with corticosteroids first but only with antibodies, it was included in this category.
  The Kaplan-Meier estimate of steroid-resistant acute rejection within the first 6 months following transplantation is reported. Participants lost to follow-up or with missing outcomes were censored at their last follow up visit.
Time Frame: 6 months
Population: Full analysis set
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Alefacept
Number analyzed (Participants) | 107 | 105
percentage of participants | 7.6 [3.4 to 11.9] | 5.7 [2.0 to 9.5]
Statistical Analysis 1: Comparison: Placebo vs Alefacept; Test type: Superiority or Other; Difference = -1.9, 90% CI 2-sided [-7.6 to 3.8]

8. Secondary Outcome: Percentage of Participants With Biopsy-Confirmed Acute T-cell Mediated Rejection as Assessed by Central Review at Month 6
Description: Biopsies were graded by the central reviewer according to the Banff 97/05 updated histological classification. A biopsy confirmed acute rejection was an event of suspected acute rejection confirmed by a graft biopsy result of Banff grade ≥ 1.
  The Kaplan-Meier estimate of biopsy-confirmed acute T-cell mediated rejection within the first 6 months following transplantation is reported. Participants lost to follow-up or with missing outcomes were censored at their last follow up visit.
Time Frame: 6 months
Population: Full analysis set
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Alefacept
Number analyzed (Participants) | 107 | 105
percentage of participants | 9.6 [4.8 to 14.3] | 7.7 [3.4 to 12.0]
Statistical Analysis 1: Comparison: Placebo vs Alefacept; Test type: Superiority or Other; Difference = -1.8, 90% CI 2-sided [-8.2 to 4.6]

9. Secondary Outcome: Patient Survival
Description: Patient survival is any participant known to be alive at Month 6. The Kaplan-Meier estimate of patient survival within the first 6 months following transplantation is reported. Participants lost to follow-up were censored at the time of last assessment.
Time Frame: 6 months
Population: Full analysis set
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Alefacept
Number analyzed (Participants) | 107 | 105
percentage of participants | 97.1 [94.4 to 99.8] | 99.0 [97.3 to 100.0]
Statistical Analysis 1: Comparison: Placebo vs Alefacept; Test type: Superiority or Other; Difference = 1.9, 90% CI 2-sided [-1.3 to 5.0]

10. Secondary Outcome: Graft Survival
Description: Graft survival was defined as any participant who was known to have a functioning graft (i.e., not graft loss) at 6 months. Graft loss is defined as re-transplantation, nephrectomy, death or as dialysis ongoing at end of study or at discontinuation of the participant unless superseded by follow-up information.
  The Kaplan-Meier estimate of graft survival within the first 6 months following transplantation is reported. Participants lost to follow-up were censored at the time of last assessment.
Time Frame: 6 months
Population: Full analysis set
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Alefacept
Number analyzed (Participants) | 107 | 105
percentage of participants | 90.6 [86.0 to 95.3] | 95.2 [91.7 to 98.6]
Statistical Analysis 1: Comparison: Placebo vs Alefacept; Test type: Superiority or Other; Difference = 4.6, 90% CI 2-sided [-1.2 to 10.4]

11. Secondary Outcome: Maximum Histological Grade of All Biopsies After Local Review
Description: The grade of acute rejection was classified according to Banff 97/05 updated version. If a patient had more than 1 rejection episode, the episode with the most severe grade was used.
  Acute T-cell mediated rejection:
  * Grade IA: significant interstitial infiltration (>25% parenchyma affected) and foci of moderate tubulitis;
  * Grade IB: significant interstitial infiltration (>25% parenchyma affected) and foci of severe tubulitis;
  * Grade IIA: mild to moderate intimal arteritis;
  * Grade IIB: severe intimal arteritis comprising >25% of the luminal area;
  * Grade III: "transmural" arteritis and/or arterial fibrinoid change and necrosis of medial smooth muscle cells with accompanying lymphocyte inflammation.
  Acute antibody-mediated rejection:
  * Grade I: acute tubular necrosis-like - complement split product positive (C4d+), minimal inflammation;
  * Grade II: capillary-margination and/or thromboses, C4d+
  * Grade III: arterial - v3, C4d+.
Time Frame: 6 months
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alefacept
Number analyzed (Participants) | 107 | 105
percentage of participants
  T-Cell Mediated Rejection - No Event | 93.5 | 89.5
  T-Cell Mediated Rejection - Grade IA | 2.8 | 1.9
  T-Cell Mediated Rejection - Grade IB | 0.0 | 1.0
  T-Cell Mediated Rejection - Grade IIA | 1.9 | 4.8
  T-Cell Mediated Rejection - Grade IIB | 1.9 | 2.9
  T-Cell Mediated Rejection - Grade III | 0.0 | 0.0
  Antibody Mediated Rejection - No Event | 97.2 | 96.2
  Antibody Mediated Rejection - Grade I | 2.8 | 1.9
  Antibody Mediated Rejection - Grade II | 0.0 | 1.9
  Antibody Mediated Rejection - Grade III | 0.0 | 0.0

12. Secondary Outcome: Percentage of Participants With Anti-Lymphocyte Antibody Therapy for Treatment of Rejection at Month 6
Description: The Kaplan-Meier estimate of anti-lymphocyte antibody therapy for acute rejection (clinically-treated or biopsy-confirmed) within the first 6 months following transplantation is reported. Participants lost to follow-up or with missing outcomes were censored at their last follow-up visit.
Time Frame: 6 months
Population: Full analysis set
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Alefacept
Number analyzed (Participants) | 107 | 105
percentage of participants | 4.7 [1.3 to 8.2] | 6.7 [2.7 to 10.7]
Statistical Analysis 1: Comparison: Placebo vs Alefacept; Test type: Superiority or Other; Difference = 2.0, 90% CI 2-sided [-3.3 to 7.2]

13. Secondary Outcome: Change From Month 1 in Serum Creatinine
Time Frame: Month 1, 3, and 6
Population: Full analysis set participants with available data at Month 1 (99 and 94 participants in each treatment group respectively) and at Month 3 and Month 6 (indicated by "n").
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Placebo | Alefacept
Number analyzed (Participants) | 99 | 94
µmol/L
  Change From Month 1 to Month 3 (n=94, 88) | -5.0125 (37.97017) | -5.0830 (66.25416)
  Change From Month 1 to Month 6 (n=86, 81) | -6.1777 (41.57056) | -11.7212 (76.19852)

14. Secondary Outcome: Change From Month 1 in Glomerular Filtration Rate (GFR)
Description: The GFR was calculated using the Modification of Diet in Renal Disease (MDRD) formula.
Time Frame: Month 1, 3, and 6
Population: Full analysis set participants with available data at Month 1 (98, 93 participants respectively) and at Month 3 and Month 6 (indicated by "n").
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m²
Arm/Group | Placebo | Alefacept
Number analyzed (Participants) | 98 | 93
mL/min/1.73 m²
  Change From Month 1 to Month 3 (n=93, 87) | 3.1548 (13.59730) | 0.2889 (12.54716)
  Change From Month 1 to Month 6 (n=83, 78) | 2.4275 (15.79533) | 2.5444 (13.06726)

15. Secondary Outcome: Change From Month 1 in Creatinine Clearance
Description: The creatinine clearance was calculated according to the Cockcroft-Gault formula.
Time Frame: Month 1, 3, and 6
Population: Full analysis set participants with available data at Month 1 (90, 84) and at Month 3 and Month 6 (indicated by "n").
Measure: Mean (Standard Deviation); unit: mL/minute
Arm/Group | Placebo | Alefacept
Number analyzed (Participants) | 90 | 84
mL/minute
  Change From Month 1 to Month 3 (n=81, 79) | 3.0336 (13.97651) | -0.5849 (12.95160)
  Change From Month 1 to Month 6 (n=77, 73) | 4.5388 (17.56456) | 3.0227 (13.25005)

16. Secondary Outcome: GFR Measured by Iothalamate Clearance at Month 6
Description: GFR measured using the iothalamate clearance method and determined by a central laboratory.
Time Frame: Month 6
Population: Full analysis set participants with available data
Measure: Mean (Standard Deviation); unit: mL/minute
Arm/Group | Placebo | Alefacept
Number analyzed (Participants) | 68 | 62
mL/minute | 59.6029 (31.36836) | 55.1613 (26.46383)

17. Secondary Outcome: Percentage of Participants With Efficacy Failure at Month 6
Description: Efficacy failure is defined as death, graft loss, biopsy-confirmed acute T-cell mediated rejection assessed by local reading or lost to follow-up.
  The Kaplan-Meier estimate of efficacy failure within the first 6 months following transplantation is reported.
Time Frame: 6 months
Population: Full analysis set
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Alefacept
Number analyzed (Participants) | 107 | 105
percentage of participants | 15.0 [9.3 to 20.6] | 21.0 [14.4 to 27.5]
Statistical Analysis 1: Comparison: Placebo vs Alefacept; Test type: Superiority or Other; Slope = 6.0, 90% CI 2-sided [-2.7 to 14.6]

18. Secondary Outcome: Percentage of Participants With Delayed Graft Function
Description: Delayed graft function was defined as the requirement for dialysis within the first week post-transplant.
Time Frame: 1 week
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alefacept
Number analyzed (Participants) | 107 | 105
percentage of participants | 12.1 | 7.6
Statistical Analysis 1: Comparison: Placebo vs Alefacept; Test type: Superiority or Other; Difference = -4.5, 90% CI 2-sided [-11.2 to 2.2]

19. Secondary Outcome: Percentage of Participants With Treatment Failure at Month 6
Description: Treatment failure is defined as efficacy failure (death, graft loss, biopsy-confirmed acute T-cell mediated rejection assessed by local reading, lost to follow-up) or early discontinuation of alefacept/placebo at any time (during the 12-week administration period) for any reason. The Kaplan-Meier estimate of treatment failure within the first 6 months following transplantation is reported. Participants lost to follow-up or with missing outcomes were censored at their last follow-up visit.
Time Frame: 6 months
Population: Full analysis set
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Alefacept
Number analyzed (Participants) | 107 | 105
percentage of participants | 20.6 [14.1 to 27.0] | 25.7 [18.7 to 32.7]
Statistical Analysis 1: Comparison: Placebo vs Alefacept; Test type: Superiority or Other; Difference = 5.2, 90% CI 2-sided [-4.4 to 14.7]

20. Secondary Outcome: Number of Participants With Adverse Events
Description: Causally related was defined as adverse events (AEs) assessed by the Investigator as possibly or probably related to study drug or records where the relationship was missing.
  A serious adverse event (SAE) was any untoward medical occurrence that, at any dose:
  * Resulted in death.
  * Was life-threatening.
  * Resulted in persistent or significant disability/incapacity.
  * Resulted in congenital anomaly or birth defect.
  * Required patient hospitalization or led to prolongation of hospitalization
  * Was considered a medically important event.
  All rejections and any BK virus, Epstein Barr virus and/or cytomegalovirus infection had to be reported as an SAE
Time Frame: 6 Months
Population: Safety analysis set (all randomized participants who received at least one dose of study drug).
Measure: Number; unit: participants
Arm/Group | Placebo | Alefacept
Number analyzed (Participants) | 107 | 105
participants
  Any adverse event | 102 | 101
  AE causally related to alefacept/placebo | 36 | 41
  AE causally related to MMF | 56 | 56
  AE causally related to tacrolimus | 49 | 49
  AE causally related to steroids | 46 | 46
  Serious adverse events | 62 | 57
  SAE causally related to alefacept/placebo | 19 | 16
  SAE causally related to MMF | 19 | 21
  SAE causally related to tacrolimus | 14 | 20
  SAE causally related to steroids | 11 | 15
  AE leading to discontinuation of alefacept/placebo | 7 | 10
  AE leading to discontinuation of MMF | 8 | 6
  AE leading to discontinuation of tacrolimus | 8 | 3
  AE leading to discontinuation of steroids | 1 | 2
  Deaths | 3 | 1

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Placebo | Alefacept
Serious Adverse Events (participants affected / at risk) | 62/107 | 57/105
Other Adverse Events (participants affected / at risk) | 98/107 | 92/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=107) | Alefacept (N=105)
Cytomegalovirus infection (Infections and infestations) | 6 | 9
Pyelonephritis (Infections and infestations) | 0 | 4
Bk virus infection (Infections and infestations) | 8 | 3
Urinary tract infection (Infections and infestations) | 6 | 2
Pyelonephritis acute (Infections and infestations) | 2 | 1
Urosepsis (Infections and infestations) | 2 | 1
Cytomegalovirus viraemia (Infections and infestations) | 1 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Epstein-barr virus infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 0 | 1
Renal abscess (Infections and infestations) | 0 | 1
Wound abscess (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Polyomavirus-associated nephropathy (Infections and infestations) | 2 | 0
Septic shock (Infections and infestations) | 2 | 0
Arteriovenous fistula site infection (Infections and infestations) | 1 | 0
Erythema infectiosum (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0
Mastitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0
Renal cyst infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Renal impairment (Renal and urinary disorders) | 8 | 4
Renal failure acute (Renal and urinary disorders) | 1 | 4
Hydronephrosis (Renal and urinary disorders) | 0 | 4
Renal artery stenosis (Renal and urinary disorders) | 3 | 1
Renal haemorrhage (Renal and urinary disorders) | 1 | 1
Renal tubular necrosis (Renal and urinary disorders) | 1 | 1
Ureteric stenosis (Renal and urinary disorders) | 1 | 1
Microalbuminuria (Renal and urinary disorders) | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Renal ischaemia (Renal and urinary disorders) | 0 | 1
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 1 | 0
Renal vein thrombosis (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 8 | 8
Chronic allograft nephropathy (Injury, poisoning and procedural complications) | 0 | 1
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 1
Graft loss (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Postoperative hernia (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Thrombosis in device (Injury, poisoning and procedural complications) | 0 | 1
Graft dysfunction (Injury, poisoning and procedural complications) | 4 | 0
Transplant failure (Injury, poisoning and procedural complications) | 2 | 0
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Perinephric collection (Injury, poisoning and procedural complications) | 1 | 0
Perirenal haematoma (Injury, poisoning and procedural complications) | 1 | 0
Urinary anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0
Histology abnormal (Investigations) | 11 | 6
Blood creatinine increased (Investigations) | 4 | 1
C-reactive protein increased (Investigations) | 0 | 1
Blood creatine increased (Investigations) | 1 | 0
Haematocrit decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 4
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Duodenogastric reflux (Gastrointestinal disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Periodontitis (Gastrointestinal disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Phaeochromocytoma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Lymphocele (Vascular disorders) | 2 | 1
Circulatory collapse (Vascular disorders) | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Iliac artery stenosis (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Hyperparathyroidism tertiary (Endocrine disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 1
Oedema peripheral (General disorders) | 0 | 1
Chest pain (General disorders) | 2 | 0
Drug intolerance (General disorders) | 1 | 0
Face oedema (General disorders) | 1 | 0
Generalised oedema (General disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 | 1
Epididymitis (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 1 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=107) | Alefacept (N=105)
Anaemia (Blood and lymphatic system disorders) | 54 | 42
Leukopenia (Blood and lymphatic system disorders) | 15 | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 5
Tachycardia (Cardiac disorders) | 1 | 6
Abdominal pain (Gastrointestinal disorders) | 4 | 7
Abdominal pain upper (Gastrointestinal disorders) | 3 | 8
Constipation (Gastrointestinal disorders) | 20 | 19
Diarrhoea (Gastrointestinal disorders) | 29 | 25
Nausea (Gastrointestinal disorders) | 7 | 10
Vomiting (Gastrointestinal disorders) | 7 | 8
Oedema peripheral (General disorders) | 14 | 9
Pyrexia (General disorders) | 9 | 9
Urinary tract infection (Infections and infestations) | 25 | 26
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 12 | 10
Procedural pain (Injury, poisoning and procedural complications) | 6 | 3
Blood creatinine increased (Investigations) | 8 | 10
Diabetes mellitus (Metabolism and nutrition disorders) | 13 | 13
Hypercholesterolaemia (Metabolism and nutrition disorders) | 7 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 14 | 17
Hyperkalaemia (Metabolism and nutrition disorders) | 10 | 10
Hyperlipidaemia (Metabolism and nutrition disorders) | 7 | 6
Hyperuricaemia (Metabolism and nutrition disorders) | 7 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 7 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 17 | 15
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 | 7
Hypophosphataemia (Metabolism and nutrition disorders) | 8 | 2
Headache (Nervous system disorders) | 4 | 7
Tremor (Nervous system disorders) | 8 | 16
Anxiety (Psychiatric disorders) | 7 | 4
Insomnia (Psychiatric disorders) | 12 | 11
Dysuria (Renal and urinary disorders) | 7 | 4
Renal impairment (Renal and urinary disorders) | 8 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 4
Hypertension (Vascular disorders) | 19 | 25
Lymphocele (Vascular disorders) | 8 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data or 12 months after data-lock, whichever is first. Sponsor must receive a site's manuscript at least 30 days prior to publication for review and comment. Sponsor may delay the publication temporarily to seek patent protection.